CLINICAL TRIAL: NCT05348642
Title: Study to Evaluate the Effect of Pasteurized Akkermansia Muciniphila (pAkk) on Complaints Related to Irritable Bowel Syndrome
Brief Title: Study to Evaluate the Effect of Pasteurized Akkermansia Muciniphila (pAkk) on Complaints Related to IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A-Mansia Biotech S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A-M/001322-2
Record Dates: First submitted 2022-04-11; First posted 2022-04-27 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Parallel Assignment randomized, double-blind, placebo-controlled, parallel group, single center trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group receiving pasteurized Akkermansia muciniphila (Experimental): pasteurized Akkermansia muciniphila - daily oral dose
  Interventions: Dietary Supplement: pasteurized A. muciniphila
- Control group (Placebo Comparator): Control group receiving placebo, identical to verum regarding the form, size, taste, color and intake.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: pasteurized A. muciniphila — pasteurized A. muciniphila - oral daily dose
  Arms: Experimental group receiving pasteurized Akkermansia muciniphila
Dietary Supplement: placebo — Placebo = identical to verum regarding the form, size, taste, color and intake
  Arms: Control group

SUMMARY:
Double-blind, randomised, placebo-controlled study to evaluate the benefit of pasteurized Akkermansia muciniphila in reducing complaints related to irritable bowel syndrome.

Further objectives are to evaluate the beneficial potential of pAkk on any anxiety and depression complaints, as well as its safety and tolerability.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is one of the most common disorders of gut-brain interaction, globally affecting about 10% of the population. Typical predominant traits are abdominal pain and abnormal bowel habits. The use of probiotics in IBS has been continuously assessed; in recent systematic reviews and meta-analyses, single or combined probiotic strains were indicated to have beneficial effects and good tolerability in the affected population.

pAkk has recently been assessed as a safe novel food ingredient. Beneficial effects and very good tolerability of pAkk have been reported in individuals with metabolic disorders. The objective of the present clinical study - a double-blind, randomised, placebo-controlled, parallel group design, explorative pilot 12-week nutritional study, is to assess the potential of pAkk in IBS management.

The main study objective is then to evaluate the benefit of pAkk in reducing complaints related to irritable bowel syndrome. Further objectives are to evaluate the beneficial potential of pAkk on any anxiety and depression complaints, as well as its safety and tolerability. In total, 90 participants will be enrolled and will attend 4 study visits: one on site and 3 televisits.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women from 18 to 70 years old
2. Meeting Rome-IV criteria for IBS:

   Recurrent abdominal pain on average ≥1 day/ week in ≥3 months prior to study (with symptom onset ≥6 months prior to study), associated with ≥2 of the following criteria:
   * Related to defecation
   * Associated with a change in frequency of stool
   * Associated with a change in form (appearance) of stool
3. Consistent and stable body weight in the last 3 months prior to study (less than 5% self-reported change)
4. Having access to a smartphone or a computer with an internet access, either allowing a video call, and familiar with the use thereof (checked during the visit)
5. Subject's agreement to comply with study procedures, in particular:

   * to take IP as recommended
   * to avoid the use of other products which may influence the GI complaints during the study
   * to keep the habitual dietary habits, type and level of physical activity (including any specific exercise such as e.g. yoga) as well as the level of caffeine or nicotine (if any)
   * to complete the subject diary and study questionnaires
6. Women of childbearing potential:

   * commitment to use contraception methods
   * negative pregnancy testing (beta human chorionic gonadotropin test in urine)
7. Readiness not to participate in another clinical study during this study

Exclusion Criteria:

1. Self-reported known allergy or hypersensitivity to any of the components of the investigational product
2. Self-reported nocturnal GI complaints
3. Women of childbearing potential: self-reported GI complaints mainly related to menstruation
4. Self-reported lactose or fructose intolerance
5. Self-reported acute or chronic significant GI disease or digestion/absorption disorders (e.g. inflammatory bowel disease, coeliac disease, pancreatitis, disorders in digestive tract motility etc.)
6. Self-reported local anorectal problems (e.g. anal fissure, bleeding haemorrhoids)
7. Self-reported clinically significant findings in colonoscopy within the 2 years prior to study
8. Family history (immediate family) of colorectal cancer or inflammatory bowel disease; anxiety or depression requiring medication
9. Acute or chronic psychiatric disease (e.g. depression, anxiety, bipolar disorder) requiring medication
10. History and/or presence of other clinically significant condition/disorder, which per investigator's judgement could interfere with the results of the study or the safety of the subject, e.g.:

    * unstable thyroid gland disorder
    * unstable hypertension
    * unstable diabetes mellitus
    * eating disorder
    * immunodeficiency
    * relevant gynecological or urological disorder
    * any other relevant serious organ or systemic diseases (e.g. cardiovascular, liver, renal disease etc.)
11. Significant GI surgery within the last 6 months prior to or planned during the study
12. Regular medication and/or supplementation within the last month prior to and during the study:

    * antibiotics, probiotics, metformin
    * for management of IBS complaints, such as bile acid binders (e.g. cholestyramine), rifaximin, alosetron, lubiprostone, eluxadoline, linaclotide, peppermint oil
    * that could influence gastrointestinal functions (e.g. laxatives, opioids, systemic corticosteroids, anticho-linergics, anti-diarrheals etc.) as per investigator judgement
13. Regular use of psychotropic drugs (e.g. hypnotics / sedative drugs, anxiolytics, antidepressants, neuroleptics, anticonvulsants) within 3 months prior to study or adaptogens (e.g. ginseng, St. John's Wort) within 6 weeks prior to and during the study
14. Introductions of a specific diet (e.g. low carb, vegan, high-fibre, low FODMAP within last 3 months prior to and during the study
15. Women of child-bearing potential: pregnancy or nursing
16. History of or current abuse of drugs, alcohol or medication
17. Participation in another study during the last 30 days prior to and during the study
18. Any other reason for exclusion as per investigator's judgment, e.g. insufficient compliance with study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Severity Scoring System / IBS-SSS | From baseline to day 14, day 42 and day 84
  Changes at each timepoint of assessment in comparison to baseline. IBS-SSS is between 0 and 500, with a higher score meaning more severe symptoms.

SECONDARY OUTCOMES:
Irritable Bowel Syndrome-Global Improvement Scale / IBS-GIS | From baseline to day 14, day 42 and day 84
  Changes at each timepoint of assessment in comparison to baseline. The IBS-GIS is a single item assessment of overall IBS symptoms. It poses the question to study participants "How would you rate your IBS signs or symptoms over the past 7 days": Subjects respond on a scale of 1-7 where: 1 = Significantly relieved, 2 = Moderately relieved, 3 = Slightly relieved, 4 = Unchanged, 5 = Slightly worse, 6 = Moderately worse, 7 = Significantly worse.
3-day diary data on stool frequency | From baseline to day 84
  Changes at each timepoint of assessment in comparison to baseline
3-day diary data on stool consistency (Bristol Stool Form Scale / BSFS) | From baseline to day 14, day 42 and day 84
  Changes at each timepoint of assessment in comparison to baseline. The Bristol Stool Form Scale is a 7 score visual scale to measure stool consistency. (1) Separate hard lumps like nuts (difficult to pass); (2) Sausage-shaped but lumpy; (3) Like a sausage but with cracks on its surface; (4) Like a sausage or snake, smooth and soft; (5) Soft blobs with clear-cut edges (passed easily); (6) Fluffy pieces with ragged edges, a mushy stool; (7) Watery, no solid pieces, entirely liquid.
Hospital Anxiety and Depression Scale / HADS | From baseline to day 14, day 42 and day 84
  Changes at each timepoint of assessment in comparison to baseline. The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains. Patients were defined as having anxiety or depression or both if the score was 8 or more in the corresponding subscale.
SF-12: 12-item Short Form survey | From baseline to day 42 and day 84
  Changes at each timepoint of assessment in comparison to baseline. The SF-12 consists of 12 items questioned weighted and summed to provide physical and mental health scores (PCS and MCS). The two composite scores are computed using the scores on twelve questions that range from 0 to 100, with higher score indicating better health.
Global evaluation of tolerability by subject and investigator | From baseline to day 84
  Changes in comparison to baseline. 8 weeks after the baseline, the subjects and the investigator will rate the tolerability of the IP by means of a global scaled evaluation with "very good", "good", "moderate" and "poor"

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — A-Mansia Biotech
Locations (1):
- analyze & realize GmbH, Berlin, Germany